CLINICAL TRIAL: NCT06242093
Title: Effects of Kegel Exercises With and Without Whole Body Vibration on Pelvic Floor Muscle Strength, Incontinence Intensity and Quality of Life in Patients With Stress Urinary Incontinence
Brief Title: Effects of Kegel ex's With and Without WBV on PFM Strength, Incontinence Intensity, and QOL in Patients With SUI.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S22C14G92026
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Pelvic floor; Quality of life; urinary incontinence; pelvic floor disorders
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Pelvic Floor Disorders | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A WBVT and Conservative treatment (Experimental): WBVT and Conservative treatment
  * Group A will receive WBVT with conservative treatment. The treatment will be given with the frequency of 34 times/week for 25-30 minutes with the help of Galileo vibration platform.
  * Time: 3-4 Times/WEEK for 8 weeks
  Interventions: Device: whole body vibrator
- GROUP B Pelvic floor muscle training (PFMT) and conservative treatment. (Active Comparator): Pelvic floor muscle training (PFMT) and conservative treatment.
  * Group B will receive (PFMT) with conservative treatment. The PMFT group will be educated to do each exercise in 3-4 set with 15-20 repetitions and a 60-second relax between each set.
  * Time: 3-4 Times/WEEK for 8 weeks
  Interventions: Other: GROUP B Pelvic floor muscle training (PFMT) and conservative treatment.

INTERVENTIONS:
Device: whole body vibrator — • WBVT and Conservative treatment Group A will receive WBVT with conservative treatment. The treatment will be given with the frequency of 34 times/week for 25-30 minutes with the help of Galileo vibration platform
  Arms: GROUP A WBVT and Conservative treatment
Other: GROUP B Pelvic floor muscle training (PFMT) and conservative treatment. — Pelvic floor muscle training (PFMT) and conservative treatment.
  Group B will receive (PFMT) with conservative treatment. The PMFT group will be educated to do each exercise in 3-4 set with 15-20 repetitions and a 60-second relax between each set.
  Time: 3-4 Times/WEEK for 8 weeks
  Arms: GROUP B Pelvic floor muscle training (PFMT) and conservative treatment.

SUMMARY:
Urinary incontinence, characterized by involuntary loss of urine (International Continence Society), is a serious social and health issue whose incidence is increasing. Urinary incontinence refers to a condition in which urine is inadvertently excreted from the bladder to the urethra, usually due to a disability or an incapacity to control the bladder and urethral sphincter. Urinary incontinence is a common complaint in women, which can have an important influence on the quality of her life. Its prevalence is between 10% and 40%, and the most common form is stress urinary incontinence. Age, body mass index, genetic factors, pregnancy and delivery, and a history of hysterectomy, smoking, race, constipation and menopause have been considered as its risk factors.

DETAILED DESCRIPTION:
Urinary incontinence, characterized by involuntary loss of urine (International Continence Society), is a serious social and health issue whose incidence is increasing. Urinary incontinence refers to a condition in which urine is inadvertently excreted from the bladder to the urethra, usually due to a disability or an incapacity to control the bladder and urethral sphincter. Urinary incontinence is a common complaint in women, which can have an important influence on the quality of her life. Its prevalence is between 10% and 40%, and the most common form is stress urinary incontinence. Age, body mass index, genetic factors, pregnancy and delivery, and a history of hysterectomy, smoking, race, constipation and menopause have been considered as its risk factors.

A Randomized controlled trial will be conducted to determine the effects of Kegel exercises with and without whole body vibration on pelvic floor muscle strength, incontinence intensity and quality of life in patients with stress urinary incontinence. A sample size of 26 SUI women's will be taken, Data will be collected from the private clinical setups of Lahore by using IQOL, Urinary intensity questionnaire: Urinary Incontinence Questionnaires (King's Health Questionnaire (KHQ), Muscle strength: PERFECT scale and SF-36 Questionnaire. A written consent form will be taken from participants meeting inclusion criteria and will be randomly allocated into two groups of equal members. One group undergoing WBVT and Conservative treatment and other group with Pelvic floor muscle training with conservative treatment. The interventions will be provided for 30 minutes for 3-4 D/Week for 4 months. All participants in both groups will be evaluated before and after the treatment programs. Total duration of study will be 8 months after the approval of synopsis. Data will be analyzed by using SPSS 26.

KEY WORDS: Pelvic floor muscle strength, Quality of life, Stress urinary incontinence, Whole body vibration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed stress urinary incontinence (SUI)
* Age: 25-50
* Married
* Normal vaginal delivery

Exclusion Criteria:

* Pelvic inflammatory disease
* Recent operation (C-section)
* Perineal tears
* Chronic constipation
* Pelvic or genital cancer
* Medical problems such as heart disease that limited activities and cardiac pacemaker
* Neuromuscular disorders
* Lack of independent mobility and exercise therapy or WBVT contraindications

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — stress urinary incontinence after pregnancy.
Enrollment: 26 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The incontinence quality of life (QOL) questionnaire | 8 weeks
  A disease-specific questionnaire that measures incontinence-related quality of life (QoL).Format: 22 items evaluating concerns related to incontinence, which can be divided into 3 sub-scales: i.e. 1.avoidance and limiting behavior, 2. psycho-social impact, 3.social embarrassment. Scoring: Items are scored on a 5-point response scale with values ranging from 1 (extremely) to 5 (not at all). Scores are then transformed to a scale score ranging from 0-100 points, with higher scores indicating higher QoL
Urinary intensity questionnaire | 8 weeks
  urinary incontinence questionnaires (King's Health Questionnaire [KHQ]:To assess and to evaluate urinary function for patients at different levels of urinary function, related to urinary leakage problems, frequency problems, and related to retention problems. The King's Health Questionnaire (KHQ) was designed to evaluate the impact of urinary incontinence on the quality of life. (r= >0.60).
SF-36 | 8 weeks
  QoL was assessed by the validated Portuguese version of the self-reported MOS SF-36, which consists of eight subscales: (1) Physical Role Function, (2) Physical Functioning, (3) Bodily Pain, (4) General Health Perception, (5) Vitality, (6) Social Role Functioning, (7) Emotional Role functioning, and (8) Mental Health. A substantial body of research supports the reliability of the SF-36 measurements. Subscale scores range from 0 to 100, with a lower score indicating lower QoL for that subscale. SF-36 (Cronbach's alpha greater than 0.85, reliability coefficient greater than 0.75).
WHOLE BODY VIBRATION PLATFORM | 8 weeks
  The Galileo is a platform with a sagittal axle on which a teeterboard is tilted up and down (5 mm) at a variable frequency of 5-30 Hz. This movement produces mechanical oscillations with an average cycle length of about 40 msec, which is the time required to induce a natural monosynaptic stretching reflex in the respective muscle via the muscle spindle during one up and down movement.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Taufiq, PPDPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No